CLINICAL TRIAL: NCT03620227
Title: Effects of Beetroot Juice Supplementation in Response to Physical Exercise in Postmenopausal and Hypertensive Women
Brief Title: Effects of Beetroot Juice in Postmenopausal and Hypertensive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Ana Luiza Amaral Ribeiro, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CEP UFU 70104717.0.0000.5152
Record Dates: First submitted 2018-05-08; First posted 2018-08-08 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Menopause
Keywords: Combined Exercise; Beetroot juice; Women health
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The volunteers will do 2 days of intervention in random order with 7 days of wash out. In one of the days will consume 350ml of concentrated beet juice and in the other 350ml of placebo made with the juice itself denitratized by an anionic resin that does not alter taste, smell or color.
Who Masked: Participant, Investigator
Masking Description: The preparation and coding of the liquids will be performed by a third party so that the researchers and participants will not know which liquid is being consumed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Experimental): ingestion of beetroot juice before an exercise session.
  Interventions: Other: Exercise; Dietary Supplement: Beetroot juice
- Placebo (Placebo Comparator): ingestion of placebo before an exercise session.
  Interventions: Other: Exercise; Dietary Supplement: Placebo

INTERVENTIONS:
Other: Exercise — 40 minutes of aerobic exercise on a treadmill, with a fixed speed of 5.5 km/h and intensity imposed by treadmill inclination until it reaches the frequency zone between 60% and 75% of the reserve heart rate.
  Other Names: Exercise session
Dietary Supplement: Beetroot juice — Ingestion of 350ml of concentrated beetroot juice (400mg of nitrate) 100 minutes before an exercise session.
  Arms: Beetroot juice
Dietary Supplement: Placebo — Ingestion of 350ml of placebo (0mg of nitrate, with the same color, taste and smell) 100 minutes before an exercise session.
  Arms: Placebo

SUMMARY:
The decrease in estrogen in postmenopausal women leads an increase in endocrine metabolic dysfunctions, such as changes in lipid profile and blood pressure. Thus, one of the alternatives for prevention and treatment is the practice of physical exercise associated with diet containing precursors of nitric oxide (NO), which is a potent vasodilator. Therefore, this study intends to verify if supplementation of beetroot juice changes the hemodynamic and salivary markers in postmenopausal and hypertensive women. Therefore, the intervention consists of 350ml of concentrated beetroot juice or placebo, which will be ingested in fasting. After 2 hours will be carried out a session of aerobic physical exercise in treadmill and blood pressure will be measured each 15 minutes for 90 minutes after the end of the session, in addition to the 24-hour measurement that will be performed by an ABPM device. Salivary samples will be held: before the juice ingest, right after exercise, 90 minutes after and 24 hours after the end of the exercise. With the development of this study, it is expected to find blood pressure reduction and normalization of the inflammatory profile through salivary samples, after the period of supplementation associated with physical exercise practice.

DETAILED DESCRIPTION:
The intervention protocol will last 3 days. On the first day there will be the collection of anthropometric data, the signature of a consent term and delivery of the list of foods that should be avoided 24 hours before the tests and a treadmill familiarization. On the second and third day the physical intervention will be performed associated with juice or placebo supplementation. A wash out period of at least 7 days will be performed between the second and third day. The volunteers will arrive at the laboratory at 7am in the fasted state and will be rested until 07:20am and then the blood pressure (BP) measurement (collected three times, with an interval of 1 minute between measurements), collection of the saliva and the measurement of heart rate (HR). Approximately at 07:30am they will start drinking the juice and will have up to 15 minutes to consume. BP will be measured at 08:00am, 08:30am, 09:00am and 09:30am. At 9:30am a physical exercise session will begin, during which will be monitored by a cardio-frequency monitor, which will remain until 11h10am (period referring to the end of BP monitoring in the laboratory). At 10:10am the workout will be finished, and then the saliva will be collected. After this period, the volunteers can take up to 250 ml of water until 11:10am, and every 15 minutes, BP will also be measured. and at 11:10am a collection of saliva will be performed. The volunteers will have the period of 15 minutes to be hygienised, and at 11:25am the ABPM will be placed (ambulatory blood pressure monitor). The ABPM will be taken the day after the test at 10:10 am (time for the first post-exercise BP measurement), and the last collection of saliva will be carried out concurrently with the ABPM removal.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 50 and 70 years;
* Amenorrhea of at least 12 months;
* Being in the postmenopausal phase;
* Be controlled hypertension;
* Be able to practice physical exercises on cycle ergometers;
* Submit a certificate attesting to the ability to practice physical exercises.

Exclusion Criteria:

* Be uncompensated hypertensive in stages 2 and 3;
* To present a history of stroke or acute myocardial infarction;
* Be a smoker;
* To present physical problems or cardiovascular complications that prevent the performance of physical exercises.
* To present a diagnosis of Diabetes Mellitus;
* To present renal pathologies;
* To present gastrointestinal pathologies;
* Have hypersensitivity to nitrate;
* Make use of hormonal therapies.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Changes in rest Blood Pressure | Before and 15, 30, 45 and 60 minutes after exercise sessions
  After 15 minutes of total rest, Systolic, Diastolic and Mean blood pressure will be measured by automatic device 3 times with one minute between measurements.
Changes in Ambulatorial Blood Pressure | Every 15 minutes during 24 hours from 60 minutes after exercise
  All volunteers were submitted to a 24-hour Blood Pressure (BP) assessment by Ambulatorial Blood Pressure Monitoring (ABPM) 60 minutes after exercise. A device was used associated with a diary of examination to self-report of activities of daily living (sleep, work, food) or any event that could interfere abnormally with BP or device measurements. The device was always placed 7am and the measurements were made every 15 minutes from 7h to 23h and every 30 minutes from 23h to 7h. The monitoring was considered valid when it happened for a period of 24 hours. The following results were evaluated: systolic blood pressure; diastolic blood pressure, mean blood pressure and heart rate in awake, sleep and 24-hour periods.

SECONDARY OUTCOMES:
Changes in Heart Rate Variability | During the 20 minutes before and after the exercise and during the execution of the exercise.
  Heart Rate (HR) was recorded using a heart rate monitor in a beat-by-beat basis. HR was registered in a seat position for 20 min of rest. Prior to the HR Variability (HRV) analysis, the RR intervals (RRi) were visually inspected and filtered using a moving average filter. The HRV was analyzed in both time-, frequency- and nonlinear-domain. Being that for frequency-domain analysis, firstly the RRi series were interpolated at 4 Hz and then the signal linear trend component removal was performed using the smooth priors approach.
Changes in salivary oxidative stress | Before supplementation, right after, 60 minutes and 24 hour after exercise sessions
  The salivary was collected after 12-hours fasting and the total antioxidant capacity was evaluated using the Ferric-Ability of Plasma (FRAP) methodology and calculated from the standard trolox curve. The activity of the enzyme superoxide dismutase (SOD) was determined based on the auto oxidation capacity of pyrogallol and catalase activity (CAT) by monitoring the consumption of hydrogen peroxide at 240 nm. Lipid peroxidation levels were determined by the TBARS method (thiobarbituric acid reactive substances), using as standard a curve of 1,1,3,3-tetraethoxypropane (TMP). The total protein concentration was obtained by the Bradford method (BRADFORD, 1976), using bovine serum albumin (BSA) as standard. The amounts of nitric oxide (NO) were estimated by the determination of total nitrite by the Griess colorimetric method.
Changes in Ambulatorial Blood Pressure Variability | Every 15 minutes during 24 hours from 60 minutes after exercise
  Based on Systolic, Diastolic and Mean Ambulatorial Blood Pressure data, were calculated Blood Pressure Variability by: 24-hour standard deviation weighted by the time interval between consecutive readings; the mean diurnal and nocturnal deviations weighted for the duration of the daytime and nighttime interval; the average real variability weighted for the time interval between consecutive readings; the ambulatory arterial stiffness index calculated by the slope of the trend curve of the dispersion of pressure data; the morning surge that represents the dynamic daytime variation in morning pressure that tends to increase, being assessed from the point of least pressure during sleep in relation to the first two hours after waking; and nocturnal dipping, that represents the average percentage drop of sleep pressure in relation to wakefulness, and individuals with falls of 10% or more are considered dippers and below that are considered nom-dippers.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Guilherme, Phd, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided